CLINICAL TRIAL: NCT00832533
Title: INST 0814: The Response of Serum 25-Hydroxyvitamin D to Incidental Ultraviolet Light Exposure
Brief Title: The Response of Serum 25-Hydroxyvitamin D to Incidental Ultraviolet Light Exposure
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0814
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Melanoma
Keywords: Vitamin D; Serum 25-Hydroxyvitamin D; UV exposure; Ultraviolet Light Exposure; Skin Melanoma Advanced
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and Buccal Smear
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1.1 To detect reproducible variations of serum 25-hydroxyvitamin D levels throughout the course of one year in relationship to objectively measured levels of ultraviolet exposure.

1.2 To determine specific times within the year that would yield the most significant data that could be focused on in future, larger studies examining whether there are protective effects of serum vitamin D on the development of cutaneous melanoma

DETAILED DESCRIPTION:
We will conduct a pilot study to investigate the ability to generate a dose-response curve of serum 25-hydroxyvitamin D to incidental ultraviolet light exposure measured objectively with a computerized personal ultraviolet light radiation dosimeter among 10 healthy volunteers in New Mexico where the population is highly exposed to solar UV radiation. During the follow-up period we will collect solar exposure data through a self-reported sun exposure diary, in tandem with objective UV dosimeter data, and will collect blood samples for serum measurements. We will carry out clinical measurements of serum vitamin D, parathyroid hormone, and calcium and phosphorus ions. We will analyze the correlation between the vitamin D and the recorded UV exposure in order to evaluate physiological changes due to solar exposure. This pilot study is important for melanoma prevention as there is currently confusion among the public as to how much sun is needed for vitamin D production and when too much sun exposure will increase risk for developing melanoma.

Expected benefits of this study to the participants include obtaining an objective measure of daily ultraviolet exposure and vitamin D status and the possible need for supplementation. Expected benefits to society include determining a dose-response of vitamin D to ultraviolet light that will enhance our understanding of the balance between necessary and harmful ultraviolet exposure. The results generated in this pilot study could provide a scientific basis for designing a larger study to develop effective primary prevention against cutaneous malignant melanoma.

This pilot study will investigate the ability to generate a dose-response curve of serum 25-hydroxyvitamin D to incidental ultraviolet light exposure measured objectively with a computerized personal UVR dosimeter. The knowledge obtained will provide important pilot data a larger NIH grant to estimate the risk-benefit of solar exposure and serum vitamin D in the development and prevention of cutaneous melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Light-skinned volunteers (Caucasians including Hispanics with slightly darker complexion)
2. 18 years of age (5 men and 5 women)
3. Resident in the State of New Mexico
4. Indoor workers with no significant history of prolonged, excessive sun exposure
5. Willing to have a monthly blood draw
6. Willing to fill out the sun diary every day on different indoor/outdoor activities.
7. During the project time period potential pregnancy of women volunteers would change the risk category of the participants, and that is a reportable event to UNM HSC HRRC and the Clinical Trial Office.

Further explanation of the inclusion criteria:

This pilot study is intended to evaluate the dose-response associations between measured UV exposure and individual serum 25 (OH)-vitamin D levels. To date, there is little data and a great deal of mis-information about vitamin D. Caucasians have a variety of skin types and melanin production. This pilot study is unfunded and we know that there is extreme heterogeneity among Caucasians in their absorption of UVB and subsequent synthesis of vitamin D. Among our volunteers 2 participants with Hispanic ethnicity are represented as well. Darker-skinned individuals, such as African Americans, produce considerably less vitamin D, based on the bone health literature. Inclusion of African Americans will be critical in the future as we develop our understanding of the relationship between vitamin D and UV exposure. Our collaborator, Elizabeth Jacobs at the University of Arizona, is currently conducting a pilot study to evaluate UV and serum vitamin D among individuals with darker pigmentation. The motivation for our pilot study has to do with the balance between vitamin D and sun exposure as a risk-benefit assessment for the development of melanoma. Asians and African Americans do develop melanoma, but at a rate ten times less than Caucasians and it does not appear to be related to sun exposure; thus, to include them at this time would not allow us to focus on the medically-related issue.

Exclusion Criteria:

1. Diet high in oily fish (e.g. eating cod liver or sardines oil conserved products more than 2-3 times/week)
2. Oral vitamin D supplementation (over 1,000 IU/day amount)
3. Tanning bed use.
4. Existing pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2 participants with Hispanic ethnicity are represented as well. Darker-skinned individuals, such as African Americans, produce considerably less vitamin D. Inclusion of African Americans will be critical. Asians and African Americans do develop melanoma, but at a rate ten times less than Caucasians and it does not appear to be related to sun exposure; thus, to include them at this time would not allow us to focus on the medically-related issue.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To detect reproducible variations of serum 25-hydroxyvitamin D levels throughout the course of one year in relationship to objectively measured levels of ultraviolet exposure. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- Universtiy of New Mexico - Cancer Center, Albuquerque, New Mexico, United States